CLINICAL TRIAL: NCT00492622
Title: Pharmacokinetics of Immediate-Release vs. Delayed-Release Omeprazole in Patients With Heartburn Associated With Gastroparesis
Brief Title: Pharmacokinetics of Immediate-Release vs. Delayed-Release Omeprazole in Gastroparesis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 014.07
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Gastroparesis; Gastroesophageal Reflux Disease
Keywords: Gastroparesis; Gastroesophageal reflux disease; heartburn
MeSH Terms: conditions — Gastroparesis; Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate-release omeprazole release first (Experimental): subjects receive immediate release omeprazole for 7 days then delayed release for 7 days
  Interventions: Drug: Immediate-release omeprazole; Drug: Delayed-release omeprazole
- Delayed-release omeprazole first (Experimental): subjects receive delayed release omeprazole for 7 days then immediate release for 7 days
  Interventions: Drug: Immediate-release omeprazole; Drug: Delayed-release omeprazole

INTERVENTIONS:
Drug: Immediate-release omeprazole — Immediate-release omeprazole 40 mg qam for 7 days
Drug: Delayed-release omeprazole — Delayed-release omeprazole 40 mg qam for 7 days

SUMMARY:
The purpose of this study is to compare the blood drug levels of two prescribed medications, immediate-release omeprazole 40 mg powder and delayed-release omeprazole 40 mg capsule to determine which drug is better absorbed in patients with a slow stomach emptying (gastroparesis). Delayed-release omeprazole has a protective coating to prevent the drug omeprazole from being neutralized by stomach acid. Immediate-release omeprazole has sodium bicarbonate (antacid) which neutralizes the stomach acid, eliminating the need for a protective coating. Immediate-release omeprazole suspension may have a more rapid pharmacokinetic profile and greater overall drug absorption in gastroparesis.

DETAILED DESCRIPTION:
Hypothesis: Immediate-release omeprazole suspension may have a more rapid pharmacokinetic profile and greater overall drug absorption in gastroparesis. This will result in shorter time to maximal drug concentration, greater maximal concentration, and greater total area under the curve of the concentration vs. time plot.

Primary Objective: To compare the pharmacokinetics of omeprazole between immediate-release suspension and delayed-release capsules in patients with heartburn associated with gastroparesis.

Study design: randomized, open-labeled, crossover treatment for 7 days with 10-14 days washout. Pharmacokinetic studies will be performed after 7 days on study drug.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms of heartburn >2 days per week off antireflux therapy, defined by "a burning feeling rising from the stomach or lower chest up towards the neck"
* Symptoms of gastroparesis >1 month in duration, defined by nausea, vomiting, bloating, dyspepsia, early satiety, or effortless regurgitation.
* Prior abnormal 4-hour gastric emptying scan within the past 3 years

Exclusion Criteria:

* History of esophageal or gastric surgery
* Severe gastroparesis with any of the following: vomiting with dehydration requiring IV hydration, hospitalization, weight loss >10 % pre-illness weight, requiring feeding jejunostomy tubes
* Presence of gastric electrical stimulator
* Symptoms of retching with vomiting more than 2 days per week
* Diagnosis of diabetes
* Disorders of small bowel motility (such as pseudo-obstruction or dumping syndrome)
* Disorders of small bowel absorption
* Diagnosis of gastric outlet, small bowel or colon mechanical obstruction
* Diagnosis of acid hypersecretory syndrome
* Disorders affecting proton pump inhibitor metabolism (such as liver failure)
* Known allergy or side effects to proton pump inhibitor
* Non-ambulatory patients: bed-ridden, nursing home resident, etc.
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Wo, MD, Principal Investigator — University of Louisville
Locations (1):
- Digestive Health Center, University of Louisville Hospital, Louisville, Kentucky, United States

REFERENCES:
- [Result] Wo JM, Eversmann J, Mann S. Pharmacokinetic profile of immediate-release omeprazole in patients with gastro-oesophageal reflux associated with gastroparesis. Aliment Pharmacol Ther. 2010 Feb 15;31(4):516-22. doi: 10.1111/j.1365-2036.2009.04203.x. Epub 2009 Nov 19. PMID 19925497

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: All participants were randomized to receive all formulations so baseline measures are reported for all participants.
Period: Overall Study
Arm/Group | All Study Participants
Started | 12 (all subjects received the immediate release formulation)
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Time to Maximal Omeprazole Concentration (Tmax)
Description: Time to max concentration for Immediate release vs. Delayed release omeprazole
Time Frame: 10, 20, 30, 45, 60, 90, 120, 150, 180, 210, 240 and 300 min after the study drug was ingested on day 7 of treatment
Population: All subjects were included regardless of which formulation they received first.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- All Study Participants Immediate Release Arm: Immediate-release omeprazole: Immediate-release omeprazole 40 mg qam for 7 days
- All Study Subjects Delayed Release Arm: Delayed-release omeprazole: Delayed-release omeprazole 40 mg qam for 7 days
Arm/Group | All Study Participants Immediate Release Arm | All Study Subjects Delayed Release Arm
Number analyzed (Participants) | 12 | 12
minutes | 32 (11) | 97 (46)
Statistical Analysis 1: Comparison: All Study Participants Immediate Release Arm vs All Study Subjects Delayed Release Arm; Test type: Equivalence — Primary study objective was to compare the pharmacokinetics of omeprazole between IR and DR omeprazole in patients with GERD associated with gastroparesis; p < 0.01, paired t-tests — <0.01 is used for determining the level of significance

2. Primary Outcome: Maximal Concentration of Omerazole
Description: Maximal concentration of immediate-release vs. delayed-release omeprazole
Time Frame: 10, 20, 30, 45, 60, 90, 120, 150, 180, 210, 240 and 300 min after the study drug was ingested on day 7 of treatment
Population: All subjects were included, regardless of which formulation they received first.
Measure: Mean (Standard Deviation); unit: ng/mL plasma
Groups:
- All Study Participants Immediate Release Arm: Immediate-release omeprazole concentration: Immediate-release omeprazole 40 mg qam for 7 days
- All Study Subjects Delayed Release Arm: Delayed-release omeprazole concentration: Delayed-release omeprazole 40 mg qam for 7 days
Arm/Group | All Study Participants Immediate Release Arm | All Study Subjects Delayed Release Arm
Number analyzed (Participants) | 12 | 12
ng/mL plasma | 1979 (832) | 1625 (921)
Statistical Analysis 1: Comparison: All Study Participants Immediate Release Arm vs All Study Subjects Delayed Release Arm; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; P<0.05 was used as the level of significance with ANOVA for this endpoint

3. Primary Outcome: Area Under the Curve for Omeprazole Plasma Concentration
Description: The area under the curve for omeprazole concentration-time curve for immediate release and delayed release omeprazole.
Time Frame: 0 to 5 hrs after the study drug was ingested on treatment day 7
Population: the AUC for each formulation were combined regardless of order given
Measure: Mean (Standard Deviation); unit: mg*h/mL
Arm/Group | All Study Participants Immediate Release Arm | All Study Subjects Delayed Release Arm
Number analyzed (Participants) | 12 | 12
mg*h/mL | 3842 (1618) | 3745 (2386)
Statistical Analysis 1: Comparison: All Study Participants Immediate Release Arm vs All Study Subjects Delayed Release Arm; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.95, ANOVA — An analysis of variance model was used to compare AUC between IR and DR omeprazole using the natural logarithmic transformation. The model included the following factors: treatment, period, sequence and patient nested within the sequence

ADVERSE EVENTS:
Groups:
- Immediate Release Fomeprazole: subjects received immediate release for 7 days then delayed release for 7 days
  Immediate-release omeprazole: Immediate-release omeprazole 40 mg qam for 7 days
- Delayed Release Omeprazole: subjects receive delayed release for 7 days then immediate release for 7 days
  Delayed-release omeprazole: Delayed-release omeprazole 40 mg qam for 7 days
Arm/Group | Immediate Release Fomeprazole | Delayed Release Omeprazole
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes